CLINICAL TRIAL: NCT05804968
Title: Exploring Feasibility, Acceptability, and Effectiveness of a Digital HIV Onward Disclosure Intervention, in People Living With HIV of Sub-Saharan African Ethnicity.
Brief Title: Exploring a Digital HIV Onward Disclosure Intervention, in People Living With HIV of Sub-Saharan African Ethnicity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Holloway University (Other)
Collaborators: Barts & The London NHS Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Megan Westhead, Trainee Clinical Psychologist, Royal Holloway University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Record Dates: First submitted 2023-02-20; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Hiv
Keywords: HIV; Single Case Experimental Design; Self Disclosure; Onward Disclosure; Digital Intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital HIV self disclosure intervention (Experimental): This study will develop a digital HIV onward disclosure intervention, drawing from the HEADSUP manual (Evangeli et al., 2020), which consists of four modules, including a HIV disclosure planning component. Participants will be asked to be involved in this study for 11 weeks, consisting of three weeks baseline, four weeks intervention and four weeks follow up.
  A single case experimental design will be used to explore HIV disclosure intention, HIV disclosure behaviour, HIV disclosure motivation, general wellbeing and mood via daily and weekly measures throughout baseline, intervention and follow up phases. All these measures will be completed online via a secure qualtrics network.
  Participants will further be asked to complete a participant experiences questionnaire to explore how they found this digital intervention. This project will recruit a diverse sample of Sub-Saharan Africa adults living with HIV and residing in the U.K.
  Interventions: Other: Digital HIV Self Disclosure Intervention

INTERVENTIONS:
Other: Digital HIV Self Disclosure Intervention — This project will develop a digital HIV disclosure intervention, drawing from the HEADSUP manual (Evangeli et al., 2020), which consists of four modules, including a HIV disclosure planning component. A SCED will be used to explore HIV disclosure intention, amongst other variables throughout baseline, intervention and follow up phases. Participants will further be asked to complete a participant experiences questionnaire to explore how they found the digital intervention and assess acceptability. This project will recruit a diverse sample of Sub-Saharan Africa adults living with HIV and residing in the U.K.

SUMMARY:
Research has shown that people living with HIV struggle to disclose their HIV status to others, (a process known as self-disclosure or onward disclosure) due to associated challenges, including fear of discrimination from others. However, there are a range of potentially positive outcomes associated with self-disclosure, such as increased medication adherence, improved wellbeing, and greater social support. Consequently, people living with HIV should be adequately supported, if they wish to disclose.

This study intends to develop and assess a digital HIV disclosure intervention, based on an existing non-digital intervention, for Sub-Saharan African adults, living with HIV and residing in the U.K. Participants will be followed pre, during and post intervention, with various measures being collected throughout, including HIV disclosure behaviour, HIV disclosure intention, HIV disclosure motivation, general wellbeing and mood. Upon follow up, participants will also be asked to complete a questionnaire regarding their personal experiences of this digital intervention. It is hypothesised that this digital HIV self disclosure intervention may lead to increases in HIV disclosure intention, amongst other secondary variables. Statistical and visual analysis will allow outcomes of this intervention to be summarised and will hopefully lead to implications and suggestions for future digital HIV disclosure interventions, supporting those living with HIV to manage the self-disclosure process effectively.

DETAILED DESCRIPTION:
Aims:

This study aims to develop a digital HIV disclosure intervention (based on the HEADS-UP intervention), for Sub-Saharan African adults living in the UK, and to test this through a Single Case Experimental Design (SCED). Research questions include: Is this intervention effective in increasing people's intention to disclose their HIV status? Is this intervention acceptable for Sub Saharan African adults, living in the UK? Is this digital disclosure intervention feasible?

Design:

A single case experimental design (SCED) will be used to explore this digital HIV disclosure intervention. Nine participants will be allocated to a three week baseline phase, four week intervention phase and four week follow up phase.

Morley's assessment, measurement funnel design will be implemented for this research project, whereby measures are taken throughout baseline, intervention and follow up (Morley, 1996). Mood will be measured via a Visual Analogue Scale, daily, for each participant throughout baseline, intervention and follow up, this will be a target measure. Weekly measures will include a 1 item disclosure behaviour question, a 1 item disclosure intention question and 3 items concerning disclosure motivation, being a 1 item question concerning positive cognitions/affect, a 1 item question concerning negative cognitions/affect and a 1 item question concerning self-efficacy, all will be target measures. The full Adolescent HIV Disclosure Cognition and Affect Scale (Evangeli, 2017) and a formal standardised wellbeing measure being the WEMBWBS (Tennant et al, 2007) will be administered twice throughout the study, being pre-baseline and post follow up, these will be the standard/global measures.

This design has been chosen as it allows cases to be studied individually and in detail, whilst maintaining a level of experimental control (Morley, 1996).Furthermore, the study design allows an effect size to be established, making it comparable to results of studies using other designs (Shadish et al., 2014). This along with visual analyses will be used to provide conclusions that can be attributed to the intervention (cause and effect can be established from this design). Furthermore, SCED is appropriate for this heterogeneous client group as it allows participants to act as their own control.

During the intervention phase participants will be asked to complete a four module digital HIV disclosure intervention, each module should take around an hour to complete and a module will be sent once every week and participants will have a week to complete this. All participants will complete a three week follow up phase. This will help to show whether immediate intervention gains are maintained, and or/or capture delayed intervention gains; analyses of trend within this phase will show changes in outcome measures.

Recruitment and Setting:

The current study will recruit adults of Sub-Saharan African origin, participants will be recruited from two London based specialist HIV-services, Infection and Immunity HIV services, Royal London Hospital (Barts Health NHS Trust) and 10 Hammersmith Broadway (Chelsea and Westminster Hospital NHS Foundation Trust).

Eligible adults who are receiving medical care from these HIV services will be identified and provided with information about the study by their clinicians at regular clinic appointments. These clients will be asked if they are interested in the study and if they are willing for their details to be passed on and to be contacted by the CI. Once participants register interest, the CI will contact them via their preferred means.

When participants are contacted by the CI, they will be presented with a digital participant information sheet to read over and will be encouraged to ask any questions. They will be given sufficient time to think about the study and if they would like to participate will need to sign a consent form, which will likely be sent electronically.

Participants:

The aim is to recruit 9 participants, although this may appear a relatively small number, this is adequate due to the in-depth nature of SCED's and the high level of participant commitment required throughout each phase, due to the requirement to complete daily and weekly measures (Dallery et al., 2013). Furthermore, the number of participants was chosen according to the requirements of effect replication needed for this design, as well as pragmatically through reviewing sample sizes used in previous SCEDs. A minimum of three effect replications are required to demonstrate experimental control, across either participants, behaviours or settings (Horner et al., 2005), so a minimum of three participants are needed. Previous SECDS to evaluate technology based health interventions have recruited 4 participants (Raiff et al, 2010).

Due to the time commitment needed for the study, it may be that up to four participants drop out. In this event, and if within the overall study time frame, more participants will be recruited to yield a final sample of nine.

Completion of the digital HIV disclosure intervention and all administering of questionnaires and contact with potential and consenting participants will be conducted remotely either over the telephone or via qualtrics.

Procedure and measures:

Participants will initially be asked to complete a digital questionnaire (via Qualtrics) to collect demographic information, including gender, age, sexuality, relationship status etc.

At baseline all participants will complete a general wellbeing questionnaire being the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) and the Adolescent HIV Disclosure Cognition and Affect Scale (Evangeli, 2017), although this measure was initially created for adolescents, previous research, including the HEADSUP trial (Evangeli et al, 2020) also used the Adolescent HIV Disclosure Cognition and Affect Scale (AHDCAS: Evangeli, 2017) with an adult population (ages 18-29), and this measure was found to have high levels of Cronbach's alpha, indicating good reliability. Furthermore, a previous RHUL DClinPsy trainee Georgina Lehmann used an AHDCAS subscale to measure disclosure self-efficacy with an adult population in her thesis (The Relationship Between Onward Disclosure and Agentic and Communal Values in Young Adults with Perinatally Acquired HIV), and this measure had Cronbach's alpha of 0.74, indicating good reliability. Furthermore, no alternative multi-item comprehensive, yet, brief scale is appropriate for my study and the items within the AHDCAS do not specifically relate to adolescents and seem appropriate items for adult use also.

All participants will be allocated to the baseline phase for three weeks and during this period they will complete daily and weekly measures including a daily measure of mood, being a single item visual analogue scale. Participants will be presented with a digital visual analogue mood scale, requiring them to rate their present mood by marking a line drawn across the scale, the left edge representing 'worst' mood and right edge, 'best' mood. Visual analogue mood scales have been shown to be a valid and reliable instrument for measuring mood (Luria, 1975). The weekly measures will include a HIV self disclosure intention question being 'How much do you agree with the following statement about telling people who do not know your status that you are HIV positive?" - "I intend to tell someone new about my HIV status in the next 6 months". Responses will be on a 5-point Likert scale from strongly disagree to strongly agree. Participants will also complete a HIV disclosure behaviour measure weekly being 'Have you shared your HIV status with anyone new over the past week?'. Participants will also be asked three questions, weekly, relating to HIV disclosure motivation, with one question relating to positive cognitions/affect, one question relating to negative cognitions/affect and one question relating to self efficacy (a person's own confidence in their ability to exert control over one's own disclosure motivations and behaviours associated with HIV disclosure). All these measures will be taken remotely via qualtrics and participants will be reminded to complete these via text message from the CI.

Once the baseline phase has commenced, the intervention phase will begin, this will last for four weeks for all participants. The digital HIV disclosure intervention consists of four modules, therefore each self-guided module will be sent to participants at the beginning of the week (Monday) and participants will be asked to complete it by the end of the week (Sunday), participants will be sent the next module, even if they have not completed the previous one. During the intervention phase daily and weekly measures will continue to be taken including a daily measure of mood and weekly measures of HIV disclosure intention, HIV disclosure behaviours and HIV disclosure motivation, as mentioned above in more detail. There will also be a measure of adherence to the intervention gathered, collected through participant self-reports.

Once the intervention phase has ended, the follow up phase will begin, this will last a total of four weeks for each participant. During this phase participants will continue to complete daily measure of mood, and weekly measures concerning HIV disclosure intention, HIV disclosure behaviour and HIV disclosure motivation. At the end of the follow up phase participants will be asked to complete the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) and the Adolescent HIV Disclosure Cognition and Affect Scale again, in order to compare pre and post study outcomes. Lastly participants will be asked to complete a Participant Experiences Questionnaire, which will be a short questionnaire to assess acceptability and feasibility of the intervention. This questionnaire will draw from the HEADS-UP acceptability questionnaire with some modified questions. One example of a question is "How likely would you be to recommend the intervention to a friend in the same situation as you", with answers ranging on a 7-point Likert scale from 'Very unlikely' to 'Very likely'. Again all measures will be completed remotely via qualtrics.

Broad Timeframe:

Recruitment is expected to begin in July/August 2023. Potential participants will be approached by their clinical care team. All clinical staff will have an understanding of the inclusion and exclusion criteria of the study. Service users who may be suitable will be introduced to the study and asked if they would like to find out more information from the CI. A meeting with the CI will be arranged to take place within the week, this will be remotely either via telephone or video call to reduce participants travel and time burden. During this meeting the CI will provide the potential participant with full information and answer any questions. Informed consent will be attained, ideally at least 24 hours after this meeting so that participants can think about this decision, and so that the CI can see that the client is able to retain the information provided to them and make an informed decision. The outcome measures will be explained to the participant by the CI, and participants will be shown how to complete them online via qualtrics. Once consent is given participants will begin the baseline phase on the agreed data. They will be expected to participate in this study for a total of 11 week (3 weeks baseline, 4 weeks intervention and 4 weeks follow up) and will be asked to complete daily and weekly measures, alongside the HIV digital intervention and a post follow up participant experiences questionnaire. The research is expected to have been fully collected by May 2024 and the final report will be prepared by June 2024. Once results are analysed, participants will be able to see them if they so wish to. They will be provided in an accessible format.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as HIV positive.
* Be an adult between the ages of 18 and 65 years old.
* Identify ethnically as sub-Saharan African.
* Have a good level of spoken and written English to ensure full engagement with the digital HIV disclosure intervention.
* Have access to a smart phone or laptop to complete the digital intervention and the associated measures.

Exclusion Criteria:

* Evidence of significant imminent risk of harm to self, or others, as identified from other professionals and clinical notes.
* Evidence of acute and very severe mental distress, as identified from other professionals.
* Significant ongoing safeguarding issues, as identified in participants' clinical notes or by the participant themselves.
* Have previously participated in the HEADS-UP HIV disclosure intervention trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HIV Disclosure Intention after 11 weeks | Up to 11 weeks
  Measured by a single item disclosure intention question.
Acceptability of Intervention | After study completion
  Measured by a participant experiences questionnaire, concerning how they found the digital HIV disclosure intervention.
Feasibility of the Intervention | Up to 11 weeks
  Measured by recruitment and retention rates and adherence rates to the modules of the digital HIV disclosure intervention.

SECONDARY OUTCOMES:
Change from baseline mood after 11 weeks | Up to 11 weeks
  Measured by a single item visual analogue scale.Participants will be presented with a digital visual analogue mood scale, requiring them to rate their present mood by marking a line drawn across the scale, the left edge representing 'worst' mood and right edge, 'best' mood.
Change from baseline HIV Self Disclosure Behaviour after 11 weeks | Up to 11 weeks
  Measured by a single item disclosure behaviour question- 'Have you shared your HIV status with anyone new over the past week?'.
Change from baseline HIV Self Disclosure Motivation after 11 weeks | Up to 11 weeks
  Measured by three items including 1 question concerning positive cognitions/affect, 1 question concerning negative cognitions/affect and 1 question concerning self-efficacy.
Change from baseline Mental Wellbeing after 11 weeks | Up to 11 weeks
  The Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS), includes 14 items. Higher scores indicate greater positive mental wellbeing.
Change from baseline HIV Disclosure Cognition and Affect after 11 weeks | Up to 11 weeks
  Adolescent HIV Disclosure Cognition and Affect Scale (AHDCAS, Evangeli, 2017), includes 18 items.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Westhead, MSc, Principal Investigator — Royal Holloway University

IPD SHARING:
Plan to Share IPD: No